CLINICAL TRIAL: NCT07291336
Title: Accuracy Assessment of Dynamic Vs. Static Navigation Implant Placement Protocols (Randomized Controlled Trial)
Brief Title: Comparing Dynamic Navigation to Static Navigation in the Implant Placement
Acronym: RCT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Salma Nabil Ahmed Lotfy Mobarek, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1113
Record Dates: First submitted 2025-11-22; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adults; Dental Implant; Accuracy
Keywords: dynamic navigation; static navigation; guide; Accuracy; delayed implant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sCAIS (Active Comparator)
  Interventions: Device: Static Implant guide
- dCAIS (Experimental)
  Interventions: Device: Dynamic navigation system

INTERVENTIONS:
Device: Dynamic navigation system — Dynamic navigation system called MiniNavident
  Other Names: dCAIS
  Arms: dCAIS
Device: Static Implant guide — Tooth supported guide is prefabricated before the surgery
  Arms: sCAIS

SUMMARY:
Implant placement is preplanned by taking xrays and impressions for the mouth one group a guide is fabricated and used to guide the implant drilling all through to the implant placement the other group, no guide is fabricated, but the implant is placed by dynamic navigation through looking in a screen and checking where the implant is fully placed

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients at least 22 years old.

  * At least one missing tooth to be restored using an implant in the upper jaw from the maxillary right 2nd premolar to the maxillary left 2nd premolar.
  * At least six residual teeth in the affected jaw (5).
  * Minimum of 5 mm available bone.

Exclusion Criteria:

* Medical condition or medication that would impair bone healing.

  * Poor oral hygiene
  * Inadequate bone width or height that may need bone augmentation. 5
  * Alcohol users.
  * Smoking more than 10 cigarettes per day.
  * History of head and neck radiotherapy.
  * Pregnant females.
  * Uncontrolled hypertensive or diabetic patient.
  * Vulnerable group; prisoners, pregnant women, orphans…etc

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Deviation | Baseline, Day 0
  Deviation in Apical position, platform position and angular deviation

SECONDARY OUTCOMES:
Patient Satisfaction Questionnaire | 1 week
  Patient satisfaction from procedure
Time | Perioperative/ Periprocedural
  Operating time taken for each procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT07291336/Prot_000.pdf